CLINICAL TRIAL: NCT04629287
Title: A Randomized, Blind, Placebo-controlled,Single Andmultiple Ascending Dose Study to Assess the Safety,Tolerability, and Pharmacokinetic of KPCXM18 for Injection in Healthy Subjects
Brief Title: Safety,Tolerability, and Pharmacokinetic of KPCXM18 for Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: KPCXM18/C101; CTR20202022 (Other: National Medical Products Administration)
Record Dates: First submitted 2020-11-03; First posted 2020-11-16 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized, blind, dose-incrementing, placebo controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KPCXM18 for injection (Experimental): KPCXM18 ，freeze-dried powder,single and multiple ascending doses, Intravenous route
  Interventions: Drug: KPCXM18; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, freeze-dried powder,single and multiple ascending doses, Intravenous route
  Interventions: Drug: KPCXM18; Drug: Placebo

INTERVENTIONS:
Drug: KPCXM18 — KPCXM18,blind,freeze-dried powder,ascending doses，Intravenous route
Drug: Placebo — Placebo,blind,freeze-dried powder,ascending doses，Intravenous route

SUMMARY:
to assess the safety,Tolerability, and pharmacokinetic of KPCXM18 for injection in healthy subjects

DETAILED DESCRIPTION:
To explore the safety, tolerance and pharmacokinetic of KPCXM18 for injection in healthy subjects by intravenous administration of different doses in single and multiple administration safety, tolerance and pharmacokinetic tests, and to obtain the safe dose range of the test drugs, thus providing dose design basis for phase II clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 19 and 26 kg/m2；male body weight not less than 50.0kg,female body weight not less than 45.0kg ；
2. General physical examination and physical and chemical examination are qualified.
3. Volunteers can communicate well with the investigator, understand and comply with the relevant requirements of the study, understand and sign the informed consent；

Exclusion Criteria:

1. Any condition that might interfere with the procedures or tests in this study;
2. Drinking（more than 14 units of alcohol per week） in 6 months ;
3. Smoking (more than 10 cigarettes per day or equal amount of tobacco) within 3 months (90 days) ;
4. Have special requirements on diet, or cannot follow a unified diet ;
5. Used a clinical trial drug within 3 months prior to administration ;
6. Positive blood pregnancy test of female subjects ;
7. Subjects may not be able to complete the study for other reasons or the investigator considers that they should not be included .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with abnormal vital signs | through study completion, an average of 2 week
  To evaluate the safety KPCXM 18 for Injection with placebo after multiple intravenous dose in healthy Chinese subjects in terms of abnormal vital signs
Number of subjects with abnormal laboratory | through study completion, an average of 2 week
  To evaluate the safety KPCXM 18 for Injection with placebo after multiple intravenous dose in healthy Chinese subjects in terms of abnormal laboratory
Number of subjects with abnormal physical examination | through study completion, an average of 2 week
  To evaluate the safety KPCXM 18 for Injection with placebo after multiple intravenous dose in healthy Chinese subjects in terms of abnormal physical examination
Number of subjects with abnormal electrocardiogram | through study completion, an average of 2 week
  To evaluate the safety KPCXM 18 for Injection with placebo after multiple intravenous dose in healthy Chinese subjects in terms of abnormal electrocardiogram
Number of subjects with adverse events | through study completion, an average of 2 week
  To evaluate the safety KPCXM 18 for Injection with placebo after multiple intravenous dose in healthy Chinese subjects in terms of abnormal adverse events

SECONDARY OUTCOMES:
Pharmacokinetics of KPCXM18 in plasma: Cmax | Time Frame: Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters：Cmax of KPCXM18 after the first day administer
Pharmacokinetics of KPCXM18 in plasma: Tmax | Time Frame: Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters：Tmax of KPCXM18 after the first day administer
Pharmacokinetics of KPCXM18 in plasma: AUC0-∞ | Time Frame: Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters： AUC0-∞ of KPCXM18 after the first day administer
Pharmacokinetics of KPCXM18 in plasma:t1/2 | Time Frame: Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters： t1/2 of KPCXM18 after the
Pharmacokinetics of KPCXM18 in plasma: Cmax,ss | Time Frame: Between Day 1 to 14 days
  To characterize the pharmacokinetic parameters：Cmax,ss of KPCXM18 after the 14th day administer
Pharmacokinetics of KPCXM18 in plasma: AUC0-∞,ss | Time Frame: Between Day 1 to 14 days
  To characterize the pharmacokinetic parameters：AUC0-∞,ss of KPCXM18 after the 14th day administer
Pharmacokinetics of KPCXM18 in plasma: Tmax,ss | Time Frame: Between Day 1 to 14 days
  To characterize the pharmacokinetic parameters：Tmax,ss of KPCXM18 after the 14th day administer

CONTACTS AND LOCATIONS:
Overall Officials: yuhong huang, Prof., Principal Investigator — Second Affiliated Hospital of Tianjin University of TCM

IPD SHARING:
Plan to Share IPD: No